CLINICAL TRIAL: NCT03088995
Title: Pre-operative Screening for HIV and Viral Hepatitis B and C: Pilot Study in Stomatology
Brief Title: Pilot Study of HIV and Hepatitis B and C Screening in Surgery
Acronym: OPDEP
Status: Completed | Type: Observational
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Other Study IDs: CREPATS 006
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-03

CONDITIONS: HIV Infections; Hepatitis B; Hepatitis C
MeSH Terms: conditions — HIV Infections; Hepatitis B; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Pilot study — Pilot study of HIV and viral hepatitis B and C screening in surgery

SUMMARY:
The purpose of the OPDEP pilot study is to assess the feasibility of implementing a pre-operative HIV / HCV / HBV screening proposal for all persons over 18 years of age and refer for surgical intervention under general anesthesia in the Department of Stomatology of the Pitié-salpêtrière hospital.

Patients undergoing treatment in Stomatology have particular areas at risk for the infections we are looking for: young patients, precarious situation, drug use, migrants ...

The aim is to evaluate the conditions for a generalization of screening in the framework of the preoperative assessment.

DETAILED DESCRIPTION:
The HIV epidemic is still active in France, with 7 000 to 8 000 new infections per year.There are an estimated 150,000 people living with HIV in France. Data from the hidden epidemic show that:

* approximately 30,000 patients are unaware of their HIV status
* that the Ile de France area accounts for 44% of new infections. For over 20 years, the patient-initiated HIV counseling and testing system has helped thousands of people to know about their HIV status, but coverage for counseling and testing low. In 2007, WHO and UNAIDS published guidance on provider-initiated HIV counseling and testing in health facilities to improve acceptance and access to prevention, treatment And care.

It is in this context that, in France, the National Plan for the Fight against AIDS and Sexually Transmitted Infections (STI) 2010-2014 recommended strengthening the screening strategies, making it its Public Health dimension, Reintegrating into an overall preventive approach. The expected benefits of routine screening would thus be individual as well as collective: routine screening could be a means of controlling infection by modifying risk behaviors, it could be a preventive tool by allowing earlier diagnosis Of the disease, it could be associated with an evolution of the management and the prognosis of the infection by allowing the initiation of an antiretroviral treatment in the acute phase of the infection. In 2011, the Ministry of Health systematized the screening proposal to the entire population, considering this strategy as cost-effective with a direct individual benefit and a Public Health benefit by reducing the number of transmission. In this Plan, health authorities recommend that hospital doctors and city general practitioners prescribe HIV testing much more widely than they do, while targeting persons belonging to an identified risk group and those Low "apparent" risk.

Screening remains a critical problem in the management with 20-30% of patients diagnosed at a late stage (CD4 <200 / mm3).

According to the Institute of Health Watch, about 100 000 hepatitis C viral patients are undiagnosed in France with differences in prevalence according to sex and age.

For hepatitis B, 55% of chronic carriers of the HBs antigen do not know their status, ie about 160 000 people in France.

The recommendations of the 2014 expert report (Dhumeaux report) have changed screening not only because of the high proportion of patients not aware of their serological status, but also of recent advances in the treatment of these two infections.

For hepatitis C, the availability of more effective, better tolerated and shorter treatments reinforces the need to screen, monitor and eventually treat the patient according to treatment recommendations.

The expert report proposes to:

* Continue targeted screening based on the risk factors for contamination (drug addiction, sexual exposure, originating from countries with high endemicity, etc.) and to inform the general population and general practitioners
* Expand the screening strategies to the following populations: men aged 18 to 60, pregnant women from the first prenatal consultation, by regularly evaluating these strategies
* Associate in all cases the research of the three viruses HBV, HCV and HIV, taking into account the epidemiological similarities, the possibility and the interest of grouped tests.

The success of screening programs depends on a number of fundamental principles including:

* Targeted disease must be associated with high morbidity and mortality
* The screening test must be safe, acceptable and inexpensive
* Effective treatment must be available These 3 principles are just for HIV, viral hepatitis B and C. HIV is associated with an increase in morbidity and mortality in the absence of antiretroviral treatment. The serological test is safe, acceptable and inexpensive. Antiretroviral therapy is available, and in 2015, French and international guidelines provide universal treatment regardless of the stage of infection.

Hepatitis C is associated with increased morbidity and mortality in the absence of treatment. The disease progresses to cirrhosis, hepatocellular carcinoma and terminal liver disease, which are responsible for high morbidity and may also be associated with severe extrahepatic manifestations. A serological test is available, safe, acceptable and inexpensive. The antiviral treatment is available with new strategies and new molecules allowing a cure in more than 95% of the patients according to the stage of the disease.

Hepatitis B is associated with increased morbidity and mortality in the absence of treatment. The serological test is safe, acceptable and inexpensive. The disease progresses to cirrhosis, hepatocellular carcinoma and terminal liver disease, which are responsible for high morbidity. Antiviral treatment is available and helps control long-term infection.

These 3 pathologies, targets of our screening, respond to these fundamental principles.

The investigators hypothesize that pre-operative screening will increase the number of HIV-positive people screened and decrease the number of people who have been treated late for their HIV, HBV and / or HCV infection. The persons detected in this way could be taken care of in optimal care channels more precisely. Moreover, knowledge of their seropositivity should modify their behavior and favor the rupture of the transmission. The proposed methodology is based on the development of a screening strategy for HIV and B and C viral hepatitis by serology, which is systematically proposed by the anesthesiologist to all persons over the age of 18 who are undergoing surgery under anesthesia In Stomatology. This study is based on the formalization of close and effective functional links between the Department of Infectious Diseases and Tropical Diseases, the Department of Stomatology and the Laboratory of Virology.

ELIGIBILITY:
Inclusion Criteria:

* men and women

  -> 18 years
* address for surgical intervention under general anesthesia in the Department of Stomatology of Pitié-Salpêtrière.
* have given their oral consent during the consultation of anesthesia.

Exclusion Criteria:

* refusal of screening
* any patient already known to be HIV-positive / HBV / HCV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-operative screening for HIV and viral hepatitis B and C: Pilot study in stomatology, Pitie salpetriere hospital.
  This study is part of a study to evaluate routine care. Screening for HIV and viral hepatitis B and C is a common clinical practice, and the populations on which it is practiced are both populations with risk behaviors and the general population. The evaluation of the strategy for scaling up HIV testing in healthcare facilities is broadly based, including a report by the National AIDS Council and the HAS and WHO recommendations that call for enlargement Of the existing screening offer.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Measure of HIV infection to assess the conditions for a generalization of screening in the Framework of the preoperative assessment | 12 months
  Measure of HIV infection assessed by serology using ARCHITECT Ag/Ac VIH Combo kit
Measure of viral hepatitis B infection to assess the conditions for a generalization of screening in the Framework of the preoperative assessment | 12 months
  Measure of viral hepatitis B infection assessed by serology using ARCHITECT AgHBs qualitative II kit
Measure of viral hepatitis C infection to assess the conditions for a generalization of screening in the Framework of the preoperative assessment | 12 months
  Measure of viral hepatitis C infection assessed by serology using ARCHITECT Anti-HCV kit

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pourcher-martinez, MD, PhD, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (1):
- Yasmine Dudoit, Paris, France

IPD SHARING:
Plan to Share IPD: No